CLINICAL TRIAL: NCT03862391
Title: Evaluation of the Effects of Low Flow Anesthesia on Pain and Agitation in Patients After Recovery
Brief Title: Does Low Flow Anesthesia Reduce Postanaesthetic Emergence Agitation?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Gürkan Demir, Assistant Physician, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Sakarya School of Medicine
Record Dates: First submitted 2019-02-15; First posted 2019-03-05 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Agitated; State, Acute Reaction to Stress
Keywords: postanesthesia agitation; general anesthesia; low-flow anesthesia
MeSH Terms: conditions — Psychomotor Agitation; Stress Disorders, Traumatic, Acute | interventions — Analgesics; Antiemetics

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postsurgical Pain (Active Comparator): pain is defined as unpleasant sensation that can range from mild, localized discomfort to agony.
  Interventions: Drug: Analgesics
- Postanesthesia nausea and vomiting (Active Comparator): nausea defined as feeling of sickness or discomfort in the stomach that may come with an urge to vomit.
  Interventions: Drug: Antiemetics

INTERVENTIONS:
Drug: Analgesics — while patients are in the PACU after general anesthesia, if patients' VAS scores are higher than 3, we will give them 50 mg of deksketoprofen as analgesic.
  Arms: Postsurgical Pain
Drug: Antiemetics — while patients are in the PACU after general anesthesia, if patient' Nausea and vomiting scores are higher than 1, we will give them 4 mg of ondansetron
  Arms: Postanesthesia nausea and vomiting

SUMMARY:
In this study, the investigators aimed to compare postanesthetic agitation in patients undergoing laparotomic gynecological surgery under general anesthesia using sevoflurane at a fresh gas flow rate of 2 L / min with fresh gas flow rate of 0.5 L / min.

DETAILED DESCRIPTION:
Emergence agitation is a temporary state of mental anxiety that occurs during general anesthesia recovery. It is characterized by emergence agitation, hallucination, excitation, delusion and confusion. Increased hemorrhage due to hypertension may cause serious complications such as injury to the surgical site, patients' self-removal of surgical drains and catheters, and self-extubation. Due to these, emergence agitation results need for additional treatment, psychological stress and increased medical workload for patients and their families.

Emergence agitation after general anesthesia in adult patients was reported up to 20%. However, the ratios are very wide.

In our operating room, the investigators observed that patients with low flow anesthesia were less agitated in the recovery phase than patients with normal flow anesthesia. In our researches, the investigators have not found any studies on the agitation values of patients who underwent low flow anesthesia in the literature.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1 and 2, underwent gynicological laparotomic surgery under general anesthesia, followed up in PACU(postoperative care unit)

Exclusion Criteria:

* ASA 3 or 4, mental retardation, psychiatric disease, history of malignant hyperthermia in patient or her family, neurological disease, morbid obesity, history of asthma and follow-up in the intensive care unit.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — we have performed our study with laparotomic gynecological surgeries
Enrollment: 60 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Postanesthetic emergence agitation | 30 minutes after general anesthesia recovery
  Emergence agitation is a temporary state of mental anxiety that occurs during general anesthesia recovery. It is characterized by emergence agitation, hallucination, excitation, delusion and confusion.
  Emergence agitation is defined as the Riker sedation-agitation scale (SAS) score of 5 or more at any time in the PACU.
  Riker sedation-agitation scale:
  7 point is 'Dangerous agitation' 6 point is 'very agitated' 5 point is 'agitated' 4 point is 'calm and cooperative' 3 point is 'sedated' 2 point is 'very sedated'
  1 point is 'unarousable'

SECONDARY OUTCOMES:
postanesthetic nausea and vomiting | 30 minutes after general anesthesia recovery
  The Nausea-Vomiting score will also assess and 4 mg of Ondansetron iv will be administered to those who had a score of 2 or more.
  The Nausea-Vomiting score:
  0 point: no nausea or vomiting
  1. point: the patient has moderate nausea for less than 15 minutes
  2. point: the patient has nausea for more than 15 minutes
  3. point: the patient has retching or vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Ali Fuat Erdem, Professor, Study Director — Lecturer
Locations (1):
- Sakarya University Training and Research Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No